CLINICAL TRIAL: NCT03084068
Title: A Prospective, Randomized Controlled Trial for Rotator Cuff Repair - Efficacy of Supraspinatus Tendon Repair Using a Human Dehydrated Umbilical Cord Patch
Brief Title: Use of Human Dehydrated Umbilical Cord Allograft in Supraspinatus Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACORT001
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Shoulder Injury; Shoulder Sprain; Supraspinatus Tear
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human umbilical cord allograft (Experimental): Open Rotator Cuff Repair patched with human dehydrated umbilical cord allograft
  Interventions: Other: Human dehydrated umbilical cord allograft
- Placebo Control (Placebo Comparator): Open Rotator Cuff Repair with standard suture repair
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Human dehydrated umbilical cord allograft — human dehydrated umbilical cord allograft
  Arms: Human umbilical cord allograft
Other: Placebo — Open rotator cuff surgery with standard suture repair
  Arms: Placebo Control

SUMMARY:
To determine the effectiveness of human dehydrated umbilical cord allograft in standard open rotator cuff repair as assessed by the American Shoulder and Elbow Surgeons (ASES) score 12 months post-op.

ELIGIBILITY:
Inclusion Criteria:

1. MRI confirmed diagnosis of a full thickness supraspinatus tendon tear necessitating surgical intervention (rotator cuff repair)
2. Subject is male or female age 18 or older
3. Subject is willing and able to provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study

Exclusion Criteria:

Subjects who meet ANY of the following criteria will be excluded from the study:

1. Shoulder pain primarily attributed to any of the following:

   1. Ligament rupture due to use of fluoroquinolones
   2. Capsular tear
   3. Fracture of the humeral head
   4. Inflammation of the joint or surrounding tissue (i.e. osteoarthritis, bursitis)
   5. Neuropathic, radiating pain from conditions resulting in damage or inflammation of the nerve
   6. Previous history of autoimmune connective tissue disorders (i.e. rheumatoid arthritis, systemic lupus erythematosus)
2. Known history of poor compliance with medical treatments
3. Subject has bilateral supraspinatus tendon tear
4. Subject has signs and symptoms of an active infection of the shoulder joint
5. Retraction of the supraspinatus tendon exceeding 1.5 cm in length
6. Subject has additional injuries requiring further surgical intervention to the ipsilateral arm
7. Subject has had previous surgery in the target arm within the past 6 months prior to treatment or plans to have surgery other than Rotator Cuff Repair in the target arm within 180 days of treatment
8. Subjects currently receiving radiation therapy or chemotherapy
9. Subjects has used an investigational drug, device or biologic within 12 weeks prior to treatment
10. Subjects who are pregnant at enrollment or are planning to become pregnant within 180 days of treatment
11. Subject has any significant medical condition(s) that, in the opinion of the Investigator, would interfere with protocol evaluation and participation
12. Allergy or known sensitivity to aminoglycoside antibiotics such as gentamicin sulfate and/or streptomycin sulfate
13. Workers' compensation patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
ASES score | 12 months
  The primary endpoint of the study is the number of subjects achieving a 20% increase from baseline in the overall ASES score at 12 months post-op.

SECONDARY OUTCOMES:
Constant Murley Score | 12 months
  Comparison of Constant scores between the two groups at each study time point
Shoulder range of motion | 12 months
  Assessment of the change in the range of motion of the shoulder joint for both treatment groups at each study time point.
VAS Pain scores | 12 months
  Change in patient reported pain from baseline
Incidence of tendon re-tear | 12 months
  Incidence of supraspinatus tendon re-tear in the two treatment groups as assessed by review of MRI scans by independent radiologists
Incidence of adverse events | 12 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Mason, MD, Study Director — MiMedx Group, Inc.
Locations (1):
- Hand & UpperEx Center, Wexford, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No